CLINICAL TRIAL: NCT00022048
Title: Safety and Efficacy Trial of Bevacizumab: Anti-VEGF Humanized Monoclonal Antibody (NSC 704865) Therapy for Myelodysplastic Syndrome (MDS)
Brief Title: Bevacizumab in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SUMC-MDA-ID-01152; CDR0000068778 (Registry Identifier: PDQ (Physician Data Query)); MDA-ID-01152; NCI-2771
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2004-10

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Bevacizumab

INTERVENTIONS:
Biological: bevacizumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them.

PURPOSE: This phase I/II trial is to see if bevacizumab works in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the hematologic responses, including changes in hemoglobin levels, neutrophil counts, platelet counts, and percentage of bone marrow blasts, in patients with myelodysplastic syndrome treated with bevacizumab.
* Determine the toxic effects of this regimen in these patients.
* Determine the tolerance in patients treated with this regimen.
* Determine bone marrow cytogenetic responses in patients treated with this regimen.
* Determine bone marrow microvessel density in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to International Prognostic Scoring System risk status (low (low or intermediate-1) vs high (intermediate-2 or high)).

Patients receive bevacizumab IV over 30-90 minutes. Treatment repeats every 2 weeks for 4-6 months in the absence of disease progression or unacceptable toxicity.

Patients are followed at weeks 1, 3, 5, 7, and 9.

PROJECTED ACCRUAL: A total of 16-25 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed myelodysplastic syndrome (MDS)

  * Refractory anemia (RA)
  * RA with excess blasts (RAEB)
  * RAEB in transformation
  * RA with ringed sideroblasts
  * Non-proliferative chronic myelomonocytic leukemia (WBC less than 12,000/mm^3)
* At least 1 of the following cytopenias:

  * Untransfused hemoglobin no greater than 10.0 g/dL and/or red cell transfusion dependent
  * Absolute neutrophil count no greater than 1,800/mm^3 (neutropenia)
  * Platelet count no greater than 100,000/mm^3 (thrombocytopenia)
* No secondary MDS
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2
* Karnofsky 60-100%

Life expectancy:

* More than 4 months

Hematopoietic:

* See Disease Characteristics
* Platelet count at least 20,000/mm^3
* No hemorrhagic illness within the past 3 weeks
* No hemolysis
* No iron deficiency
* No active blood loss

Hepatic:

* AST and ALT no greater than 2.5 times upper limit of normal (ULN)
* Bilirubin no greater than 2.0 mg/dL
* INR less than 2.0
* PTT less than 1.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL
* No renal dysfunction requiring dialysis within the past 6 months
* No nephrotic syndrome within the past 6 months

Cardiovascular:

* No myocardial infraction within the past 6 months
* No severe or unstable angina within the past 6 months
* No severe peripheral vascular disease (ischemic rest pain, non-healing wound or ulcer, or tissue loss) within the past 6 months
* No uncontrolled hypertension within the past 6 months
* No transient ischemic attack within the past 6 months
* No cerebrovascular accident within the past 6 months
* No deep venous or arterial thrombosis
* No coronary artery disease
* No symptomatic congestive heart failure (New York Heart Association class II-IV heart disease)
* No cardiac arrhythmia
* No vascular illness within the past 3 weeks

Pulmonary:

* No pulmonary embolism

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy except localized squamous cell or basal cell skin cancer

  * Prior cured malignancy allowed
* No trauma within the past 3 weeks
* No significant inflammatory disease within the past 3 weeks
* No serious non-healing wound, ulcer, or bone fracture
* No hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* No other active severe disease
* No infection
* No psychiatric illness or social situation that would preclude study compliance
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior allogeneic bone marrow transplantation
* At least 30 days since prior biologic response modifiers
* At least 30 days since prior hematopoietic growth factors
* At least 30 days since prior thalidomide
* No concurrent thalidomide
* No other concurrent biologic response modifiers
* No concurrent hematopoietic growth factors (including epoetin alfa)
* Concurrent filgrastim (G-CSF) for febrile neutropenia allowed
* Concurrent transfusions allowed

Chemotherapy:

* At least 30 days since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* No concurrent corticosteroid therapy (more than 10 mg/day of prednisone or equivalent steroid dose) except for pre-medication for transfusions

Radiotherapy:

* At least 30 days since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since prior surgery (including biopsy of visceral organ)

Other:

* At least 10 days since prior anticoagulants
* No concurrent cytotoxic agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Greenberg, MD, Study Chair — Stanford University
Locations (3):
- United States (3):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - University of Texas - MD Anderson Cancer Center, Houston, Texas